CLINICAL TRIAL: NCT03966079
Title: Single-dose rtPA Thrombolysis Endovascular Treatment of Pulmonary Embolism With Right Ventricular Dysfunction:a Pilot Study
Brief Title: Thrombolysis Endovascular Treatment of Pulmonary Embolism
Acronym: STEP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BeijingTCGH
Record Dates: First submitted 2019-05-20; First posted 2019-05-29 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Pulmonary Embolism; Acute Pulmonary Embolism
Keywords: Acute Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Intervention Model Description: Prospective Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention arm (Experimental): Patients receive 20 mg of single-dose recombinant tissue plasminogen activator delivered through the catheter
  Interventions: Drug: recombinant tissue plasminogen activator

INTERVENTIONS:
Drug: recombinant tissue plasminogen activator — Patients receive 20 mg of single-dose recombinant tissue plasminogen activator delivered through the catheter
  Other Names: rtPA

SUMMARY:
To assess the efficacy and safety of endovascular thrombolysis of pulmonary embolism with right ventricular dysfunction with single-dose rtPA

DETAILED DESCRIPTION:
The patients with right ventricular dysfunction who are diagnosed by CT pulmonary angiography will receive 20 mg of single-dose recombinant tissue plasminogen activator delivered through the in this study. The Change of RV to LV Diameter Ratio,Rate of death,rate of major bleeding,pulmonary embolism recurrence at 1month will be reviewed to assess the efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* CT evidence of proximal PE
* Age ≥ 18 years
* Pulmonary embolism symptom duration ≤14 days
* Massive PE (syncope, systemic arterial hypotension, cardiogenic shock, or resuscitated cardiac arrest) OR Submassive PE (RV diameter-to-LV diameter ≥ 0.9 on contrast-enhanced chest CT)

Exclusion Criteria:

* Age <18 years
* PE symptom duration >14 days
* Stroke or transient ischemic attack (TIA), head trauma, or other active intracranial or intraspinal disease within one year
* Recent (within one month) or active bleeding from a major organ
* Pregnancy
* Chronic pulmonary hypertension or severe chronic obstructive pulmonary disease
* Administration of thrombolytic agents within the previous 3 days
* Life expectancy < 30 days
* Any other condition that the investigator feels would place the patient at increased risk if the investigational therapy is initiated
* Inability to follow protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Change of RV to LV Diameter Ratio | baseline and 30days after baseline
  Determine whether single-dose rtpa catheter-directed thrombolysis decrease the ratio of right ventricular (RV)-to-left ventricular (LV) diameter within 1month in patients with right ventricular dysfunction

SECONDARY OUTCOMES:
Rate of death | 30days
Rate of major Bleeding | 30days
Pulmonary embolism recurrence | 30days

CONTACTS AND LOCATIONS:
Overall Officials: Wu weiwei, doctor, Study Director — Director of department
Locations (1):
- Beijing Tsinghua Chang Gung Hospital, Beijing, Beijing Municipality, China